CLINICAL TRIAL: NCT06366724
Title: LIFT: Life Improvement Trial
Acronym: LIFT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Open Medicine Foundation (Unknown)
Responsible Party: Principal Investigator, David Systrom, Principal Investigator; Director, Dyspnea Center; Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P000087
Record Dates: First submitted 2024-03-20; First posted 2024-04-16 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: ME/CFS; Long COVID; PASC
Keywords: Chronic fatigue; Mestinon; Low Dose Naltrexone; Orthostatic Intolerance; Post exertional malaise; Cognitive Impairment; Long COVID
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Post-Acute COVID-19 Syndrome; Orthostatic Intolerance; Cognitive Dysfunction | interventions — Pyridostigmine Bromide; Naltrexone

STUDY DESIGN:
Intervention Model Description: Randomized factorial group double-blinded placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Mass General Brigham Investigational Drug Services (IDS) will be responsible for randomizing the four arms. The rest of the study staff and collaborators will be blinded as well as the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Pyridostigmine/LDN (Active Comparator): Pyridostigmine will be taken as liquid suspension three times a day, scaling up from 20mg (1.67mL) to 60mg (5mL) (180mg/day). Low dose naltrexone will be taken as liquid suspension once a day, scaling up from 1.5mL to 4.5mL (4.5mg/day).
  Interventions: Drug: Pyridostigmine; Drug: Low-Dose Naltrexone
- Pyridostigmine/Placebo (Active Comparator): Pyridostigmine will be taken as liquid suspension three times a day, scaling up from 20mg (1.67mL) to 60mg (5mL) (180mg/day). Placebo will be taken as liquid suspension once a day, scaling up from 1.5mL to 4.5mL.
  Interventions: Drug: Pyridostigmine; Other: Placebo
- Placebo/LDN (Active Comparator): Placebo will be taken as liquid suspension three times a day, scaling up from 1.67mL to 5mL. Low dose naltrexone will be taken as liquid suspension once a day, scaling up from 1.5mL to 4.5mL (4.5mg/day).
  Interventions: Drug: Low-Dose Naltrexone; Other: Placebo
- Placebo/Placebo (Placebo Comparator): Placebo will be taken as liquid suspension three times a day, scaling up from 1.67mL to 5mL. Placebo will be taken as liquid suspension once a day, scaling up from 1.5mL to 4.5mL .
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pyridostigmine — Pyridostigmine timeline:
  Weeks 0-2: 20mg TID (1.67 mL TID)
  Weeks 2-4: 40mg TID (3.33 mL TID)
  Weeks 5-13: 60mg TID (5mL TID)
  Other Names: Mestinon
  Arms: Pyridostigmine/LDN; Pyridostigmine/Placebo
Drug: Low-Dose Naltrexone — LDN timeline:
  Weeks 0-2: 1.5mg QD (1.5mL QD)
  Weeks 2-4: 3.0mg QD (3.0mL QD)
  Weeks 5-13: 4.5mg QD (4.5mL QD)
  Other Names: LDN
  Arms: Placebo/LDN; Pyridostigmine/LDN
Other: Placebo — Placebo timeline:
  Weeks 0-2: 20mg TID (1.67mL TID)/1.5mg QD (1.5mL QD)
  Weeks 2-4: 40mg TID (3.33mL TID)/3.0mg QD (3.0mL QD)
  Weeks 5-13: 60mg TID (5mL TID)/4.5mg QD (4.5mL QD)
  Arms: Placebo/LDN; Placebo/Placebo; Pyridostigmine/Placebo

SUMMARY:
The LIFT will be conducted at Brigham and Women's Hospital (BWH) of Harvard Medical School, focusing on the effect of Pyridostigmine (Mestinon) and Low-Dose Naltrexone (LDN) in subjects aged 18-70 meeting the Canadian consensus criteria (CCC) for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) as well as having specifically Orthostatic Intolerance (OI). Long COVID (LC) subjects will also be included if they meet CCC and have OI.

This double-blind, placebo-controlled study will involve 160 participants randomized into one of four possible groups: Pyridostigmine/LDN (40), Pyridostigmine/Placebo (40), LDN/Placebo (40), Placebo/Placebo (40). The dose of Pyridostigmine will be carefully titrated from 30mg to 60mg three times a day, and the dose of LDN will be titrated from 1.5 mg to 4.5 mg once daily.

The trial includes a scale-back plan, allowing participants to reduce their dosage if they experience intolerance symptoms, with adjustments made during weekly visits. This plan provides a personalized approach to medication tolerance, ensuring participant's safety and comfort throughout the trial.

The time commitment for the participant is approximately three (3) months, and during this time, there will be three (3) in-person visits to BWH and four (4) virtual visits. Study procedures will include two (2) submaximum cardiopulmonary exercise tests, questionnaires (virtually completed), and blood and urine collection. We will be recruiting from the BWH Dyspnea Clinic as well as the Open Medicine Foundation (OMF) StudyME Registry and anticipate the entire trial will take two (2) years to complete.

The LIFT represents a significant endeavor to improve treatment options for ME/CFS patients and contribute to the broader understanding of this debilitating condition.

ELIGIBILITY:
Inclusion Criteria:

1. Meet National Academy of Medicine Criteria, Canadian Consensus Criteria (See appendix), and demonstrate orthostatic intolerance for diagnosis of ME/CFS
2. Participant is ≥ 18 and ≤ 70 years of age at screening, inclusive.
3. The onset of symptoms prior to December 2023.
4. Female participant is not pregnant and at least 1 of the following conditions apply:

   1. Not a woman of childbearing potential
   2. Woman of childbearing potential who agrees to follow the contraceptive guidance. from the time of informed consent.
5. Participant agrees and can adhere to the study requirements for the length of the study.
6. Participant has a body mass index (BMI) range of 17 to 40 kg/m2, inclusive.
7. Participant agrees not to participate in another interventional study while participating in the present study.
8. Participant has a functioning smart phone to download and run the DANA Brain Vital Mobile Application.

Exclusion Criteria:

1. Pregnant, planning to become pregnant, or breastfeeding.
2. Any use of opioid medications within 30 days of screening.
3. Positive urine test for opioids
4. History of alcohol, opioid or other substance misuse
5. Participation in another interventional clinical trial in the last 30 days or planned during the trial period.
6. Allergy to medication components
7. Participant has any condition which, in the investigator's opinion, makes the participant unsuitable for study participation.
8. Participant has diabetes mellitus (type 1 or 2).
9. Participant has undergone an inpatient hospitalization within the 30 days prior to the randomization or has a planned hospitalization or a surgical procedure during the study, which may affect the study assessments, in the opinion of the investigator.
10. Participant has clinically significant respiratory disease (such as chronic obstructive pulmonary disease, cystic fibrosis, severe asthma, lung infections including tuberculosis, sarcoidosis, thoracic endometriosis, pulmonary fibrosis, and lung cancers) and/or cardiac disease (medical history or current clinical findings)
11. Participant has an active malignancy or any other cancer.
12. Participant has initiated an exercise regimen within 4 weeks prior to randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Functional Capacity | 15 weeks
  Change in the total FUNCAP55 questionnaire score
  The FUNCAP55 is a questionnaire developed to assess the functional capacity of patients. Each question is answered on a 6-point scale. The greater the score, the better the functioning.
Physiologic Response - Oxygen Uptake Efficiency Slope (OUES) | 13 weeks
  Changes in % of predicted oxygen uptake efficiency slope (OUES) between baseline and follow-up measured during a non-invasive cardiopulmonary exercise test (CPET)
Physiologic Response - Oxygen Utilization (VO2) | 13 weeks
  Changes in % of predicted extrapolated peak oxygen utilization (extrapolated max VO2) between baseline and follow-up measured during a submaximum CPET
Physiologic Response - Heart Rate Recovery (HRR) | 13 weeks
  Changes in 1-min heart rate recovery (HRR) in beats per minute (bpm) between baseline and follow-up measured during a submaximum CPET

SECONDARY OUTCOMES:
Post-Exertional Malaise | 15 weeks
  Change in DePaul Symptom Questionnaire-1 (DSQ1) score
  The questionnaire lists 5 symptoms that are scored based on frequency and severity. Each question is answered on a 4-point scale. The greater the score, the greater the frequency and severity of the symptom.
PROMIS-29-Pain | 15 weeks
  Change in PROMIS-29 questionnaire score
  Reflected as combination of the "pain interference" (0 to 5) and "pain intensity" (0 to 10) sections of the questionnaire will be secondary outcomes. The greater the score, the greater the pain experienced.
Daily Activity | 15 weeks
  Change in daily steps (steps/day) measured using Garmin Vivosmart 5
Heart Rate Variability | 15 weeks
  Change in heart rate variability (HRV) defined as the specific change in time (ms) between successive heart beats. All collected via Garmin VivoSmart5
Blood Oxygen | 15 weeks
  Change in blood oxygen saturation (%) measured with Garmin VivoSmart 5
Resting Heart Rate | 15 weeks
  Change in resting heart rate (bpm) using Garmin VivoSmart 5
DANA Brain Vital-Simple Reaction Time (SRT) | 15 Weeks
  Change in time (ms) required to recognize the presence of an object and tap the object
DANA Brain Vital-Procedural Reaction Time (PRT) | 15 weeks
  Change in time (ms) required to recognize 1 of 4 numbers and tap 1 of 2 buttons
DANA Brain Vital-Memory Search (MS) | 15 weeks
  Change in time (ms) required to recognize letters that have previously been memorized

CONTACTS AND LOCATIONS:
Overall Officials: David Systrom, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification(text, tables, figures, and appendices) will be available for researchers who provide a methodologically sound proposal to achieve aims in the approved proposal.
Supporting Information: SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals should be directed to jsquires1@bwh.harvard.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- See also: MGB Rally - LIFT — https://rally.massgeneralbrigham.org/study/lift_life_improvement_trial__